CLINICAL TRIAL: NCT06576323
Title: An Intervention Mapping Approach to Closing the Gap in Maternal OUD and Infant NAS Care
Brief Title: An Intervention Mapping Approach to Closing the Gap in Maternal OUD and Infant NAS Care (SUPPORT)
Acronym: SUPPORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R21DA058815 (NIH)
Record Dates: First submitted 2024-08-06; First posted 2024-08-28 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Opioid Use Disorder; Neonatal Abstinence Syndrome
MeSH Terms: conditions — Opioid-Related Disorders; Neonatal Abstinence Syndrome | interventions — Prescriptions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Case Series (Other): In Aim 3, all recruited participants will receive the intervention.
  Interventions: Behavioral: An implementation model for co-located Medications for Opioid Use Disorder (MOUD) prescription in the NICU

INTERVENTIONS:
Behavioral: An implementation model for co-located Medications for Opioid Use Disorder (MOUD) prescription in the NICU — We will use implementation mapping to develop a suite of implementation strategies to deliver evidence-based MOUD prescription to mothers attending the bedside of their infants hospitalized in the NICU. The intervention itself is buprenorphine induction and treatment, however the model for delivery is not yet developed, consistent with the need for results from Aim 1 to inform the approach used to develop the implementation model in Aim 2.

SUMMARY:
The purpose of this study is to address the gap in maternal OUD treatment and infant neonatal opioid withdrawal syndrome care. The research team will develop a treatment model and a set of strategies to provide evidence-based OUD treatment to postpartum mothers in NICUs.

First, the investigators will conduct a needs assessment via in-depth qualitative interviews with NICU mothers and clinicians. Then, with the expertise of the advisory board, the the researchers will create a protocol for implementing maternal OUD treatment at the NICU bedside. The researchers will then implement the protocol in two partner NICUs and evaluate the acceptability and feasibility to patients, providers, and clinical, and administrative leaders.

The goal of this research study is to integrate maternal mental health and substance abuse treatment in pediatric settings and to refine, test, and examine the acceptability and feasibility of applying the adapted model.

DETAILED DESCRIPTION:
The increasing prevalence of pregnant and postpartum women affected by Opioid Use Disorder (OUD) in the US is highlighted by the growing number of babies referred to the NICU for Neonatal Abstinence Syndrome after birth. Despite recent advances in integrating mental health and substance abuse treatment into adult healthcare settings, no current treatment options exist to integrate maternal OUD treatment and referrals into the pediatric care setting making it unlikely that mothers will be able to access care. In order to preserve the dyadic bond, improve maternal functioning, and provide a more stable environment for the infant after discharge from the NICU, the researchers now embark on a study utilizing steps from intervention mapping to identify facilitators and barriers to integrated maternal OUD treatment and referral in the NICU, adapt existing evidence-based models of co-located OUD care to the NICU setting, and test the feasibility and acceptability of the new model. In Aim 1, the researchers will collect qualitative data via in-depth interviews with 32 NICU providers, social workers, administrators, and parents to determine barriers and facilitators to offering bedside buprenorphine induction and treatment. In Aim 2, the researchers will convene an advisory board to review data collected in Aim 1 and to develop a plan for implementing buprenorphine initiation into the study's unique setting to address the issue- the provision of adult focused OUD care in a pediatric care setting. Aim 2 does not constitute Human Subjects research. The primary outcome of Aim 2 will be a suite of implementation strategies to pilot test in Aim 3. Aim 3 is a pilot case series implementation trial where the researchers will test the adapted intervention to determine feasibility and acceptability to both providers and patients. As this is a case series the investigators propose to recruit 10 participants from each of the two partner NICUs for a total enrollment of N= 20 in Aim 3. A formal sample size calculation was not performed as there is no data on which to a base a formal sample size calculation. For pilot studies with an expected medium standardized effect size, a case number of N= 15 per group has been recommended for pilot studies preceding a possible main study with a power of 90%. The investigators plan to recruit 20 participants to account for possible attrition. The researchers are not necessarily powered to detect an effect. Participants will not be randomized to condition; all NICU mothers meeting inclusion criteria during the study timeline for Aim 3 will be invited to participate in Aim 3. The outcomes of acceptability and feasibility will be measured through questionnaires, interviews, and treatment initiation and retention statistics.

ELIGIBILITY:
Inclusion Criteria for Interview Participants in Aim 1:

* Participants should be healthcare providers working within UPHS, who generally treat perinatal women or any individuals with OUD; for the purposes of this study, provider refers to a Medical Doctor (MD) or Doctor of Osteopathy (DO), Advanced Practice Practitioner, Nurse, or Social Worker.
* Participants should provide direct care to NICU patients and/or their mothers
* Participants should be proficient in English language
* Participants should have access to a computer with internet connectivity or phone

Inclusion Criteria for Mothers in Aim 1:

* Participants should be biological mothers of children hospitalized in the UPHS NICU for NAS
* Participants should be diagnosed with opioid use disorder

Inclusion Criteria for Clinicians in Aim 3:

* See above for inclusion criteria for interview participants.
* We will use this same criteria to recruit new participants for Aim 3 if the same stakeholder interviewees are unavailable at the time of Aim 3.

Inclusion Criteria for Mothers in Aim 3:

* Participants should be biological mothers of a child hospitalized in either of the two UPHS NICU for NAS (either HUP or PAH)
* Participants should be no more than 4 weeks postpartum
* Participants should have an Opioid Use Disorder than is currently untreated with medication assisted treatment or buprenorphine

Exclusion Criteria for Interview Participants in Aim 1:

- None

Exclusion Criteria for Mothers in Aim 1:

- None

Exclusion Criteria for Clinicians in Aim 3:

- None

Exclusion Criteria for Mothers in Aim 3:

- Active suicidal ideation, or other severe psychopathology that must be addressed before effective MOUD can be prescribed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Qualitative Interview for NICU Providers | Time 1 (baseline)
  In-depth qualitative interview focused on providers' attitudes and knowledge about barriers and facilitators of buprenorphine induction for mothers in the NICU. This interview will be guided by the Consolidated Framework for Implementation Research to query about barriers and facilitators of MOUD provision in the NICU, with the primary goal of identifying contextual determinants of co-located care.
Qualitative Interview for Parents | Time 1 (baseline)
  In-dept qualitative interview focused on mothers' attitudes about receiving MOUD in the NICU while caring for their hospitalized infant. This interview will be guided by the Consolidated Framework for Implementation Research to query about what would make this more attractive, feasible, and engagement more likely.
Feasibility of Intervention Measure | Up to 9 months
  A 4-item,psychometrically-validated measure that indexes the extent to which stakeholders perceive an implementation strategy is feasible.
Acceptability of Intervention Measure | Up to 9 months
  A 4-item,psychometrically-validated measure that indexes the extent to which stakeholders perceive an implementation strategy is acceptable.
Recruitment and Retention Statistics | Up to 1 year.
  The proportion of mothers of babies in the NICU who agree to receive MOUD in the NICU (Time 2; T2), who remain in care for the duration of their baby's stay (Time 3; T3), and length of time they remain in outpatient treatment after treatment (Time 4; T4).

OTHER OUTCOMES:
Demographics survey | Time 1 (baseline)
  Brief questionnaire about provider and parent demographic (e.g., age, gender) and professional characteristics (e.g., provider role, years of experience, level of training), and work setting

CONTACTS AND LOCATIONS:
Overall Officials: Sara Kornfield, PhD, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Center for Women's Behavioral Wellness, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hirai AH, Ko JY, Owens PL, Stocks C, Patrick SW. Neonatal Abstinence Syndrome and Maternal Opioid-Related Diagnoses in the US, 2010-2017. JAMA. 2021 Jan 12;325(2):146-155. doi: 10.1001/jama.2020.24991. PMID 33433576
- [Background] Winkelman TNA, Villapiano N, Kozhimannil KB, Davis MM, Patrick SW. Incidence and Costs of Neonatal Abstinence Syndrome Among Infants With Medicaid: 2004-2014. Pediatrics. 2018 Apr;141(4):e20173520. doi: 10.1542/peds.2017-3520. PMID 29572288
- [Background] Ray-Griffith S, Tharp E, Coker JL, Catlin D, Knight B, Stowe ZN. Buprenorphine Medication for Opioid Use Disorder: A Study of Factors Associated With Postpartum Treatment Retention. Am J Addict. 2021 Jan;30(1):43-48. doi: 10.1111/ajad.13084. Epub 2020 Jul 16. PMID 32673447
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Becker-Haimes EM, Mandell DS, Fishman J, Williams NJ, Wolk CB, Wislocki K, Reich D, Schaechter T, Brady M, Maples NJ, Creed TA. Assessing Causal Pathways and Targets of Implementation Variability for EBP use (Project ACTIVE): a study protocol. Implement Sci Commun. 2021 Dec 20;2(1):144. doi: 10.1186/s43058-021-00245-3. PMID 34930483
- [Background] Fernandez ME, Ten Hoor GA, van Lieshout S, Rodriguez SA, Beidas RS, Parcel G, Ruiter RAC, Markham CM, Kok G. Implementation Mapping: Using Intervention Mapping to Develop Implementation Strategies. Front Public Health. 2019 Jun 18;7:158. doi: 10.3389/fpubh.2019.00158. eCollection 2019. PMID 31275915
- [Background] Committee Opinion No. 711: Opioid Use and Opioid Use Disorder in Pregnancy. Obstet Gynecol. 2017 Aug;130(2):e81-e94. doi: 10.1097/AOG.0000000000002235. PMID 28742676
- [Background] Ko JY, Patrick SW, Tong VT, Patel R, Lind JN, Barfield WD. Incidence of Neonatal Abstinence Syndrome - 28 States, 1999-2013. MMWR Morb Mortal Wkly Rep. 2016 Aug 12;65(31):799-802. doi: 10.15585/mmwr.mm6531a2. PMID 27513154
- [Background] McQueen K, Murphy-Oikonen J. Neonatal Abstinence Syndrome. N Engl J Med. 2016 Dec 22;375(25):2468-2479. doi: 10.1056/NEJMra1600879. No abstract available. PMID 28002715
- [Background] Patrick SW, Schumacher RE, Benneyworth BD, Krans EE, McAllister JM, Davis MM. Neonatal abstinence syndrome and associated health care expenditures: United States, 2000-2009. JAMA. 2012 May 9;307(18):1934-40. doi: 10.1001/jama.2012.3951. Epub 2012 Apr 30. PMID 22546608
- [Background] Tolia VN, Patrick SW, Bennett MM, Murthy K, Sousa J, Smith PB, Clark RH, Spitzer AR. Increasing incidence of the neonatal abstinence syndrome in U.S. neonatal ICUs. N Engl J Med. 2015 May 28;372(22):2118-26. doi: 10.1056/NEJMsa1500439. Epub 2015 Apr 26. PMID 25913111
- [Background] Substance Abuse and Mental Health Services Administration (US); Office of the Surgeon General (US). Facing Addiction in America: The Surgeon General's Spotlight on Opioids [Internet]. Washington (DC): US Department of Health and Human Services; 2018 Sep. Available from http://www.ncbi.nlm.nih.gov/books/NBK538436/ PMID 30860690
- [Background] Ko JY, Tong VT, Haight SC, Terplan M, Snead C, Schulkin J. Obstetrician-gynecologists' practice patterns related to opioid use during pregnancy and postpartum-United States, 2017. J Perinatol. 2020 Mar;40(3):412-421. doi: 10.1038/s41372-019-0535-2. Epub 2019 Oct 15. PMID 31616051
- [Background] Seehusen DA, Baldwin LM, Runkle GP, Clark G. Are family physicians appropriately screening for postpartum depression? J Am Board Fam Pract. 2005 Mar-Apr;18(2):104-12. doi: 10.3122/jabfm.18.2.104. PMID 15798139
- [Background] Olin SS, McCord M, Stein REK, Kerker BD, Weiss D, Hoagwood KE, Horwitz SM. Beyond Screening: A Stepped Care Pathway for Managing Postpartum Depression in Pediatric Settings. J Womens Health (Larchmt). 2017 Sep;26(9):966-975. doi: 10.1089/jwh.2016.6089. Epub 2017 Apr 14. PMID 28409703
- [Background] Fernandez ME, Ruiter RAC, Markham CM, Kok G. Intervention Mapping: Theory- and Evidence-Based Health Promotion Program Planning: Perspective and Examples. Front Public Health. 2019 Aug 14;7:209. doi: 10.3389/fpubh.2019.00209. eCollection 2019. PMID 31475126
- [Background] Highfield L, Hartman MA, Mullen PD, Rodriguez SA, Fernandez ME, Bartholomew LK. Intervention Mapping to Adapt Evidence-Based Interventions for Use in Practice: Increasing Mammography among African American Women. Biomed Res Int. 2015;2015:160103. doi: 10.1155/2015/160103. Epub 2015 Oct 26. PMID 26587531
- [Background] Brownson RC, Jacobs JA, Tabak RG, Hoehner CM, Stamatakis KA. Designing for dissemination among public health researchers: findings from a national survey in the United States. Am J Public Health. 2013 Sep;103(9):1693-9. doi: 10.2105/AJPH.2012.301165. Epub 2013 Jul 18. PMID 23865659
- [Background] Volpp KG, Asch DA. Make the healthy choice the easy choice: using behavioral economics to advance a culture of health. QJM. 2017 May 1;110(5):271-275. doi: 10.1093/qjmed/hcw190. PMID 27803366
- [Background] Pomerantz AS, Sayers SL. Primary care-mental health integration in healthcare in the Department of Veterans Affairs. Fam Syst Health. 2010 Jun;28(2):78-82. doi: 10.1037/a0020341. PMID 20695667
- [Background] Lomonaco-Haycraft KC, Hyer J, Tibbits B, Grote J, Stainback-Tracy K, Ulrickson C, Lieberman A, van Bekkum L, Hoffman MC. Integrated perinatal mental health care: a national model of perinatal primary care in vulnerable populations. Prim Health Care Res Dev. 2018 Jun 18;20:e77. doi: 10.1017/S1463423618000348. PMID 29911521
- [Background] Morrison J, Hasselblad M, Kleinpell R, Buie R, Ariosto D, Hardiman E, Osborn SW, Lindsell CJ; Vanderbilt Learning Healthcare System Investigators, Vanderbilt University. The Disruptive bEhavior manageMEnt ANd prevention in hospitalized patients using a behaviORal intervention team (DEMEANOR) study protocol: a pragmatic, cluster, crossover trial. Trials. 2020 May 24;21(1):417. doi: 10.1186/s13063-020-04278-2. PMID 32448331
- [Background] Stadnick NA, Brookman-Frazee L, Mandell DS, Kuelbs CL, Coleman KJ, Sahms T, Aarons GA. A mixed methods study to adapt and implement integrated mental healthcare for children with autism spectrum disorder. Pilot Feasibility Stud. 2019 Mar 28;5:51. doi: 10.1186/s40814-019-0434-5. eCollection 2019. PMID 30976456
- [Background] Beidas RS, Volpp KG, Buttenheim AN, Marcus SC, Olfson M, Pellecchia M, Stewart RE, Williams NJ, Becker-Haimes EM, Candon M, Cidav Z, Fishman J, Lieberman A, Zentgraf K, Mandell D. Transforming Mental Health Delivery Through Behavioral Economics and Implementation Science: Protocol for Three Exploratory Projects. JMIR Res Protoc. 2019 Feb 12;8(2):e12121. doi: 10.2196/12121. PMID 30747719
- [Background] Kranzler HR, Washio Y, Zindel LR, Lynch KG, Hand D, Tyndale RF, Oncken C, Schnoll R. Pregnant Smokers Receiving Opioid Agonist Therapy Have an Elevated Nicotine Metabolite Ratio: A Replication Study. Nicotine Tob Res. 2020 Oct 8;22(10):1923-1927. doi: 10.1093/ntr/ntaa066. PMID 32303761
- [Background] Kranzler HR, Washio Y, Zindel LR, Wileyto EP, Srinivas S, Hand DJ, Hoffman M, Oncken C, Schnoll RA. Placebo-controlled trial of bupropion for smoking cessation in pregnant women. Am J Obstet Gynecol MFM. 2021 Nov;3(6):100315. doi: 10.1016/j.ajogmf.2021.100315. Epub 2021 Jan 22. PMID 33493703
- [Background] Kornfield SL, Moseley M, Appleby D, McMickens CL, Sammel MD, Epperson CN. Posttraumatic Symptom Reporting and Reported Cigarette Smoking During Pregnancy. J Womens Health (Larchmt). 2017 Jun;26(6):662-669. doi: 10.1089/jwh.2016.5928. Epub 2017 Feb 21. PMID 28437216
- [Background] Kornfield SL, Geller PA, Epperson CN. Maternal Fetal Attachment, Locus of Control and Adherence to STI/HIV Prevention and Prenatal Care Promotion Behaviors in Urban Women. Int J Gynecol Obstet Reprod Med Res. 2014;1(1):11-18. PMID 25729776
- [Background] Kornfield SL, Johnson RL, Hantsoo LV, Kaminsky RB, Waller R, Sammel M, Epperson CN. Engagement in and Benefits of a Short-Term, Brief Psychotherapy Intervention for PTSD During Pregnancy. Front Psychiatry. 2022 Jun 15;13:882429. doi: 10.3389/fpsyt.2022.882429. eCollection 2022. PMID 35782453
- [Background] Kornfield SL, White LK, Waller R, Njoroge W, Barzilay R, Chaiyachati BH, Himes MM, Rodriguez Y, Riis V, Simonette K, Elovitz MA, Gur RE. Risk And Resilience Factors Influencing Postpartum Depression And Mother-Infant Bonding During COVID-19. Health Aff (Millwood). 2021 Oct;40(10):1566-1574. doi: 10.1377/hlthaff.2021.00803. PMID 34606353
- [Background] Hamm RF, Levine LD, Nelson MN, Beidas R. Implementation of a calculator to predict cesarean delivery during labor induction: a qualitative evaluation of the clinician perspective. Am J Obstet Gynecol MFM. 2021 May;3(3):100321. doi: 10.1016/j.ajogmf.2021.100321. Epub 2021 Jan 22. PMID 33493705
- [Background] Becker-Haimes EM, Wislocki K, DiDonato S, Jensen-Doss A. Predictors of Clinician-Reported Self-Efficacy in Treating Trauma-Exposed Youth. J Trauma Stress. 2022 Feb;35(1):109-119. doi: 10.1002/jts.22688. Epub 2021 May 28. PMID 34048094
- [Background] Guest, G., Bunce, A., & Johnson, L. (2006). How Many Interviews Are Enough?: An Experiment with Data Saturation and Variability. Field Methods, 18(1), 59-82. https://doi.org/10.1177/1525822X05279903
- [Background] Potthoff S, Presseau J, Sniehotta FF, Breckons M, Rylance A, Avery L. Exploring the role of competing demands and routines during the implementation of a self-management tool for type 2 diabetes: a theory-based qualitative interview study. BMC Med Inform Decis Mak. 2019 Jan 24;19(1):23. doi: 10.1186/s12911-019-0744-9. PMID 30678684
- [Background] Hays DG, Singh AA. Qualitative inquiry in clinical and educational settings. New York, NY: Guilford; 2012
- [Background] Bradley EH, Curry LA, Devers KJ. Qualitative data analysis for health services research: developing taxonomy, themes, and theory. Health Serv Res. 2007 Aug;42(4):1758-72. doi: 10.1111/j.1475-6773.2006.00684.x. PMID 17286625
- [Background] Glaser B, Strauss A. Applying Grounded Theory. The discovery of grounded theory: strategies of qualitative research. 1967. doi: 10.4324/9780203793206.
- [Background] Palinkas LA. Qualitative and mixed methods in mental health services and implementation research. J Clin Child Adolesc Psychol. 2014;43(6):851-61. doi: 10.1080/15374416.2014.910791. PMID 25350675
- [Background] Davis R, Campbell R, Hildon Z, Hobbs L, Michie S. Theories of behaviour and behaviour change across the social and behavioural sciences: a scoping review. Health Psychol Rev. 2015;9(3):323-44. doi: 10.1080/17437199.2014.941722. Epub 2014 Aug 8. PMID 25104107
- [Background] Esposito D, Heeringa J, Bradley K, Croake S, Kimmey L, Lechner A. 2015. PCORI Dissemination and Implementation Toolkit. Princeton, NJ: Mathematica Policy Research.
- [Background] Pellecchia M, Beidas RS, Mandell DS, Cannuscio CC, Dunst CJ, Stahmer AC. Parent empowerment and coaching in early intervention: study protocol for a feasibility study. Pilot Feasibility Stud. 2020 Feb 13;6:22. doi: 10.1186/s40814-020-00568-3. eCollection 2020. PMID 32082608
- [Background] Pellecchia M, Mandell DS, Nuske HJ, Azad G, Benjamin Wolk C, Maddox BB, Reisinger EM, Skriner LC, Adams DR, Stewart R, Hadley T, Beidas RS. Community-academic partnerships in implementation research. J Community Psychol. 2018 Sep;46(7):941-952. doi: 10.1002/jcop.21981. Epub 2018 Apr 6. PMID 30565736
- [Background] Stewart RE, Beidas RS, Mandell DS. Stop Calling Them Laggards: Strategies for Encouraging Nonadopters to Incorporate Evidence-Based Practices. Psychiatr Serv. 2019 Oct 1;70(10):958-960. doi: 10.1176/appi.ps.201900031. Epub 2019 Jun 27. PMID 31242831
- [Background] Stewart RE, Adams DR, Mandell DS, Nangia G, Shaffer L, Evans AC, Rubin R, Weaver S, Hadley TR, Beidas RS. Non-participants in policy efforts to promote evidence-based practices in a large behavioral health system. Implement Sci. 2017 May 25;12(1):70. doi: 10.1186/s13012-017-0598-4. PMID 28545492
- [Background] Waltz TJ, Powell BJ, Fernandez ME, Abadie B, Damschroder LJ. Choosing implementation strategies to address contextual barriers: diversity in recommendations and future directions. Implement Sci. 2019 Apr 29;14(1):42. doi: 10.1186/s13012-019-0892-4. PMID 31036028
- [Background] Newman SD, Andrews JO, Magwood GS, Jenkins C, Cox MJ, Williamson DC. Community advisory boards in community-based participatory research: a synthesis of best processes. Prev Chronic Dis. 2011 May;8(3):A70. Epub 2011 Apr 15. PMID 21477510
- [Background] Korthuis PT, McCarty D, Weimer M, Bougatsos C, Blazina I, Zakher B, Grusing S, Devine B, Chou R. Primary Care-Based Models for the Treatment of Opioid Use Disorder: A Scoping Review. Ann Intern Med. 2017 Feb 21;166(4):268-278. doi: 10.7326/M16-2149. Epub 2016 Dec 6. PMID 27919103
- [Background] Alford DP, LaBelle CT, Kretsch N, Bergeron A, Winter M, Botticelli M, Samet JH. Collaborative care of opioid-addicted patients in primary care using buprenorphine: five-year experience. Arch Intern Med. 2011 Mar 14;171(5):425-31. doi: 10.1001/archinternmed.2010.541. PMID 21403039
- [Background] LaBelle CT, Han SC, Bergeron A, Samet JH. Office-Based Opioid Treatment with Buprenorphine (OBOT-B): Statewide Implementation of the Massachusetts Collaborative Care Model in Community Health Centers. J Subst Abuse Treat. 2016 Jan;60:6-13. doi: 10.1016/j.jsat.2015.06.010. Epub 2015 Jun 26. PMID 26233698
- [Background] Rich KM, Bia J, Altice FL, Feinberg J. Integrated Models of Care for Individuals with Opioid Use Disorder: How Do We Prevent HIV and HCV? Curr HIV/AIDS Rep. 2018 Jun;15(3):266-275. doi: 10.1007/s11904-018-0396-x. PMID 29774442
- [Background] Basu S, Smith-Rohrberg D, Bruce RD, Altice FL. Models for integrating buprenorphine therapy into the primary HIV care setting. Clin Infect Dis. 2006 Mar 1;42(5):716-21. doi: 10.1086/500200. Epub 2006 Jan 24. PMID 16447120
- [Background] Johnson E. Models of care for opioid dependent pregnant women. Semin Perinatol. 2019 Apr;43(3):132-140. doi: 10.1053/j.semperi.2019.01.002. Epub 2019 Jan 14. PMID 30981471
- [Background] State of Vermont. Vermont Blueprint for Health. Blueprintforhealth.vermont.gov
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Philadelphia Department of Public Health. Prescription Opioid and Benzodiazepine Use in Philadelphia, 2017. CHART 2017;2(9):1-6